CLINICAL TRIAL: NCT01164384
Title: A Phase 1b, Single Center, Clinical Study to Investigate the Safety and Biological Responses to Baminercept in Patients With Chronic HCV Hepatitis.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Collaborators: PD Dr. rer. nat. Mathias Heikenwälder (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BamiHepC-Study
Record Dates: First submitted 2010-07-08; First posted 2010-07-16 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Chronic HCV Hepatitis C
MeSH Terms: interventions — baminercept

INTERVENTIONS:
Drug: Baminercept

SUMMARY:
Erstes Safety Trial mit Baminercept in chronischen HCV Patienten. Untersuchung des potentiell antiviralen, antiinflammatorischen Effekts sowie Modulation der hepatischen Gen-Expression.

10 Patienten, open label, 10 Wochen Therapie. Sequentielles Enrollement der ersten 4 Patienten.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: Informed consent Age 18-60 years Chronic HCV infection Non responder (to Peg-IFN alpha2/Ribavirin containing therapy) Elevated ALT Liver biopsy at screening without sings of (pre-)cirrhosis Compensated liver function Absolute neutrophil count > 1500 / mm3 at screening Hemoglobin > 10 g/dL at screening Calculated creatinine clearance of > 60 cc/min at screening Normal TSH at screening

Exclusion criteria: HBV infection Evidence for concomitant liver disease other than HCV hepatitis Evidence for a HCC Alpha-fetoprotein >20ng/ml Autoimmune Disease ANA > 1/320, documented in the last 6 months HIV 1/2 infection ALT and AST >3x ULN, alkaline phosphatase >2,5x ULN Known hypersensitivity or allergy to Baminercept Other clinically significant concomitant disease states Known or suspected non-compliance to study protocol, drug or alcohol abuse Infections other than HCV hepatitis Clinically important chest x-ray abnormality at screening Body mass index (BMI) > 30kg/m2 Concomitant systemic immunosuppressive/-modulating therapy Treatment with anticoagulants Receipt of live vaccine within 4 weeks prior to study start Symptomatic hypogammaglobulinemia with history of recurrent infections Subjects with a history of malignant disease Treatment with other investigational products or participation in an interventional clinical trial within the last 3 months Pregnancy or Breastfeeding Inability or refusal to practice a safe contraception

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2010-10; Study Completion 2013-02

PRIMARY OUTCOMES:
Sicherheit

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland